CLINICAL TRIAL: NCT05040971
Title: Efficacy and Safety of Subcutaneous Semaglutide 2.4 mg Once-weekly in Subjects With Obesity and Prediabetes
Brief Title: Research Study Looking at How Well Semaglutide Works in People Living With Obesity and Prediabetes
Acronym: STEP 10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4734; U1111-1253-1956 (Other: World Health Organization (WHO)); 2020-002939-29 (EudraCT Number)
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive subcutaneus (s.c.) semaglutide 2.4 mg once weekly for 52 weeks
  Interventions: Drug: Semaglutide 2.4 mg
- Placebo (semaglutide) (Placebo Comparator): Participants will receive subcutaneus (s.c.) placebo (semaglutide) once weekly for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 2.4 mg — Administered subcutaneously (s.c., under the skin) once weekly as well as reduced-calorie diet and increased physical activity for 52 weeks. Doses gradually increased to 2.4 mg
  Arms: Semaglutide
Drug: Placebo — Administered subcutaneously once weekly (s.c., under the skin) as well as reduced-calorie diet and increased physical activity for 52 week
  Arms: Placebo (semaglutide)

SUMMARY:
This study looks at how well a new medicine, called semaglutide, works at helping people with obesity and prediabetes.

This study will look at how much weight participants lose, and if participants can go from having blood sugar that is higher than normal (prediabetes) to having normal blood sugar.

Semaglutide is compared to a "dummy" medicine. The "dummy" medicine looks like semaglutide but has no effect on the body.

In addition to taking the medicine, participants will have talks with study staff about healthy food choices, how to be more physically active and what participants can do to lose weight.

Participants will either get semaglutide or "dummy" medicine - which treatment they get is decided by chance. Participants are 2 times as likely to get semaglutide as "dummy" medicine.

Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm.

The study will last for about 19 months. Participants have to take the study medicine every week for the first 12 months. The last 7 months participants will not take any medication.

Participants will have 14 clinic visits and 1 phone call with the study staff. At 9 of the clinic visits Participants will have blood samples taken. Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged greater than or equal to 18 years at the time of signing informed consent.
* BMI greater than or equal to 30.0 kg/m^2
* Prediabetes defined as at least one of the following:

  * HbA1c between 6.0 and 6.4 percent (42 and 47 mmol/mol) (both inclusive) as measured by central laboratory at screening.
  * FPG between 5.5 and 6.9 mmol/L (99 and 125 mg/dL) (both inclusive) as measured by central laboratory at screening.

Exclusion Criteria:

* History of type 1 or type 2 diabetes.
* Treatment with glucose-lowering agent(s) within 90 days before screening.
* HbA1c greater than or equal to 6.5 percent (greater than or equal to 48 mmol/mol) as measured by central laboratory at screening.
* FPG greater than or equal to 7.0mmol/L (126 mg/dL) as measured by central laboratory at screening.

A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records.

* Treatment with any medication for the indication of obesity within the past 90 days before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (43):
- Canada (28):
  - LMC Clin Res Inc. Calgary, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - Weight Wise Clinic, Edmonton, Alberta
  - Ocean West Research Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - LMC Diabetes & Endocrinology (Barrie), Barrie, Ontario
  - LMC ClinRsrh Inc.Brampton, Brampton, Ontario
  - LMC Clin Res Inc. Thornhill, Concord, Ontario
  - LMC Endo Ctr (Etobicoke) Ltd, Etobicoke, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Milestone Research, London, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - LMC Clinical Research Inc. Oakville, Oakville, Ontario
  - Centricity Research LMC, Toronto, Ontario
  - Toronto Sleep Institute/MedSleep, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Dr Anil K Gupta Med Prof Corp, Toronto, Ontario
  - Manna Research Mirabel, Mirabel, Quebec
  - Centre Medical Acadie, Montreal, Quebec
  - Clinique Medicine Urbaine du Quartier Latin, Inc., Montreal, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
  - Centre de recherché du CHUS, Sherbrooke, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
  - CHU de Quebec-Universite Laval, Québec
  - Institut universitaire de cardiologie, Québec
- Denmark (2):
  - Aarhus Universitetshospital Diabetes og Hormonsygdomme, Aarhus N
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
- Finland (2):
  - Obesity Research Unit, Helsinki
  - StudyCor, Jyväskylä
- Spain (3):
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Infanta Luisa, Seville
- United Kingdom (8):
  - Clifton Medical Centre, Rotherham, South Yorkshire
  - The Health Centre, Bradford-on-Avon
  - University Hospital Coventry - WISDEM Centre, Coventry
  - Claremont Medical Practice, Exmouth
  - GP Direct, Harrow
  - Guys Hospital, London
  - The Staploe Medical Centre, Soham
  - MyHealth - Strensall Health Care Centre, Strensall

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] McGowan BM, Bruun JM, Capehorn M, Pedersen SD, Pietilainen KH, Muniraju HAK, Quiroga M, Varbo A, Lau DCW; STEP 10 Study Group. Efficacy and safety of once-weekly semaglutide 2.4 mg versus placebo in people with obesity and prediabetes (STEP 10): a randomised, double-blind, placebo-controlled, multicentre phase 3 trial. Lancet Diabetes Endocrinol. 2024 Sep;12(9):631-642. doi: 10.1016/S2213-8587(24)00182-7. Epub 2024 Jul 29. PMID 39089293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 30 sites in 5 countries as follows: Canada (15 sites), Denmark (2 sites), Finland (2 sites), Spain (3 sites) and United Kingdom (8 sites).
Pre-assignment Details: The trial has a Main phase and Extension phase. Main phase: a 52-week treatment period (16 weeks of dose escalation and 36 weeks of maintenance dose). Extension phase: a 28-week off-treatment extension phase after the main phase for assessment of body weight, glycaemic and cardiovascular parameters. Participants were randomised in 2:1 ratio either to receive semaglutide 2.4 mg or placebo as an adjunct to a reduced-calorie diet and increased physical activity.
Groups:
- Semaglutide 2.4 mg: Participants received once-weekly subcutaneous (s.c) injection of 0.25 milligram (mg) Semaglutide administered using a DV3396 pen-injector followed by a fixed-dose escalation regimen, with dose increase every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week) until the maintenance dose of 2.4 mg after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg Semaglutide once weekly for an additional 36 weeks until week 52. The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
- Placebo: Participants received once-weekly subcutaneous (s.c) injection of 0.25 milligram (mg) placebo matched to 2.4 mg Semaglutide administered using a DV3396 pen-injector followed by a fixed-dose escalation regimen, with dose increase every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week) until the maintenance dose of 2.4 mg after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg placebo matched to 2.4 mg Semaglutide once weekly for an additional 36 weeks until week 52. The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 138 | 69
Full Analysis Set (FAS) | 138 | 69
Safety Analysis Set (SAS) | 138 | 69
Completed | 128 | 64
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 8 | 3
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all the randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 138 | 69 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53 (11) | 53 (11) | 53 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 47 | 147
  Male | 38 | 22 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 132 | 68 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 124 | 59 | 183
  Asian | 4 | 5 | 9
  Black or African American | 6 | 3 | 9
  Other | 4 | 1 | 5
  American Indian or Alaska Native | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (Percentage [%])
Description: Change in body weight from randomisation (week 0) to end of treatment (week 52) is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: Full analysis set (FAS) included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage (%) of body weight
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
Percentage (%) of body weight | -14.4 (7.9) | -2.7 (4.3)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority — Week 52 responses were analysed using an analysis of covariance model (ANCOVA) with randomised treatment as factor and baseline body weight as covariate; p < 0.0001, ANCOVA; Treatment difference = -11.19, 95% CI 2-sided [-12.97 to -9.42]

2. Primary Outcome: Participants With Change to Normoglycemia
Description: Number of participants in glycaemic categories, "normoglycaemia, pre-diabetes and type 2 diabetes" at Week 52 are presented. These categories were set as per the following criteria: 1) Normoglycaemia: glycosylated haemoglobin (HbA1c) lesser than (<) 6.0 percentage (%) and fasting plasma glucose (FPG) lesser than (<) 5.5 millimoles per liter (mmol/L). 2) Pre-diabetes: 6.0% lesser than or equal (≤) HbA1c lesser than (<) 6.5% or 5.5 mmol/L lesser than or equal (≤) FPG lesser than (<) 7.0 mmol/L or non-verified type 2 diabetes. 3) Type 2 diabetes: HbA1c greater than or equal (≥) 6.5% or FPG greater than or equal (≥) 7.0 mmol/L.
Time Frame: At week 52
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 127 | 64
Participants
  Normoglycemia | 103 | 9
  Pre-diabetes | 23 | 53
  Type 2 diabetes | 1 | 2
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority — Week 52 responses were analysed using a logistic regression model with randomised treatment as factor and baseline glycosylated haemoglobin (HbA1c) and fasting plasma glucose (FPG) as covariates; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 19.81, 95% CI 2-sided [8.68 to 45.21]

3. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change in glycosylated haemoglobin (HbA1c) from randomisation (week 0) to end of treatment (week 52) is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 63
Percentage of HbA1c | -0.4 (0.3) | 0.1 (0.2)

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in fasting plasma glucose (FPG) from randomisation (week 0) to end of treatment (week 52) is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 127 | 63
millimoles per liter (mmol/L) | -0.8 (0.6) | -0.3 (0.7)

5. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from randomisation (week 0) to end of treatment (week 52) is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
centimeter (cm) | -11.6 (8.7) | -2.8 (5.4)

6. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from randomisation (week 0) to end of treatment (week 52) is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
millimeters of mercury (mmHg) | -9 (13) | -1 (13)

7. Secondary Outcome: Change in Triglycerides (Millimoles Per Liter [mmol/L]) - Ratio to Baseline
Description: Change in triglycerides (measured in mmol/L) from randomisation (week 0) to end of treatment (week 52) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 126 | 62
Ratio of triglycerides | 0.80 (36.4) | 0.96 (30.6)

8. Secondary Outcome: Change in Total Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in total cholesterol (measured in mmol/L) from randomisation (week 0) to end of treatment (week 52) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 127 | 63
Ratio of total cholesterol | 0.94 (16.1) | 1.01 (15.7)

9. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in high density lipoprotein (HDL) cholesterol (measured in mmol/L) from randomisation (week 0) to end of treatment (week 52) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 119 | 61
Ratio of HDL cholesterol | 1.02 (12.4) | 0.99 (11.7)

10. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in low density lipoprotein (LDL) cholesterol (measured in mmol/L) from randomisation (week 0) to end of treatment (week 52) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 118 | 61
Ratio of LDL cholesterol | 0.93 (26.6) | 1.03 (23.6)

11. Secondary Outcome: Change in Very Low Density Lipoprotein (VLDL) Cholesterol (mmol/L) - Ratio to Baseline
Description: Change in very low density lipoprotein (VLDL) cholesterol (measured in mmol/L) from randomisation (week 0) to end of treatment (week 52) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 125 | 62
Ratio of VLDL cholesterol | 0.80 (36.5) | 0.96 (30.7)

12. Secondary Outcome: Change in Body Weight (Kilogram [Kg])
Description: as for outcome 1
Time Frame: From randomisation (week 0) to week 52
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: kilogram (Kg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
kilogram (Kg) | -15.8 (9.3) | -2.8 (5.0)

13. Secondary Outcome: Participants Achieving Body Weight Reduction Greater Than or Equal (≥) 5% (Yes/No)
Description: Participants who achieved body weight reduction greater than or equal to 5% (Yes/No) at week 52 is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: At week 52
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
Participants
  Yes | 111 | 17
  No | 18 | 49

14. Secondary Outcome: Participants Achieving Body Weight Reduction Greater Than or Equal (≥) 10% (Yes/No)
Description: Participants who achieved body weight reduction greater than or equal to 10% (Yes/No) at week 52 is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: At week 52
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
Participants
  Yes | 95 | 5
  No | 34 | 61

15. Secondary Outcome: Participants Achieving Body Weight Reduction Greater Than or Equal (≥) 15% (Yes/No)
Description: Participants who achieved body weight reduction greater than or equal to 15% (Yes/No) at week 52 is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: At week 52
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
Participants
  Yes | 62 | 1
  No | 67 | 65

16. Secondary Outcome: Participants Achieving Body Weight Reduction Greater Than or Equal (≥) 20% (Yes/No)
Description: Participants who achieved body weight reduction greater than or equal to 20% (Yes/No) at week 52 is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: At week 52
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 66
Participants
  Yes | 32 | 0
  No | 97 | 66

17. Secondary Outcome: Change in Pulse
Description: Change in pulse from randomisation (week 0) to end of treatment (week 52) is presented. The endpoint was evaluated based on the data from in-trial observation period which was defined as the time period where the participant was assessed in the main phase of the study. The 'in-trial' (main phase) observation period for a participant begins on the date of randomisation and ends at the first of the following dates (both inclusive): safety visit, withdrawal of consent, last contact with participant (for participants lost to follow-up), death.
Time Frame: From randomisation (week 0) to end of treatment (week 52)
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 128 | 66
beats per minute (bpm) | 2 (10) | 0 (7)

ADVERSE EVENTS:
Time Frame: From randomisation (week 0) to week 57
Description: All the presented adverse events (AEs) are treatment emergent adverse events (TEAEs). Treatment emergent adverse events (TEAEs): events that had onset date during on-treatment period, time period in which participants was considered exposed to trial product. Safety analysis set (SAS) during on-treatment included all participants randomly assigned to treatment who took at least one dose of study product.
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/138 | 0/69
Serious Adverse Events (participants affected / at risk) | 12/138 | 6/69
Other Adverse Events (participants affected / at risk) | 93/138 | 30/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=138) | Placebo (N=69)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Embedded device (Product Issues) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (3) | 0 (0)
Pilonidal disease (Infections and infestations) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Submandibular abscess (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=138) | Placebo (N=69)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 4 (4)
COVID-19 (Infections and infestations) | 48 (55) | 21 (21)
Constipation (Gastrointestinal disorders) | 25 (29) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (31) | 7 (7)
Dizziness (Nervous system disorders) | 7 (7) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 12 (21) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 5 (6)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (2)
Nausea (Gastrointestinal disorders) | 40 (50) | 3 (3)
Vomiting (Gastrointestinal disorders) | 16 (27) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT05040971/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT05040971/SAP_001.pdf